CLINICAL TRIAL: NCT02220972
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Effect of Perampanel on Objective and Subjective Sleep in Subjects With Insomnia and Partial Onset Seizures
Brief Title: To Evaluate the Effect of Perampanel on Objective and Subjective Sleep in Subjects With Insomnia and Partial Onset Seizures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-408
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Partial Onset Seizures; Insomnia
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Sleep Initiation and Maintenance Disorders | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: First on Perampanel with a crossover to Placebo (Experimental): Treatment Arm A will initially receive perampanel 2 mg QD titrated up to 4 mg QD and finally to 6 mg QD with a crossover to placebo.
  Interventions: Drug: Perampanel; Drug: Placebo
- Arm B: First on Placebo with a crossover to Perampanel (Experimental): Treatment Arm B will initially receive placebo with a crossover to perampanel 2 mg QD titrated up to 4 mg QD and finally to 6 mg QD.
  Interventions: Drug: Perampanel; Drug: Placebo

INTERVENTIONS:
Drug: Perampanel
Drug: Placebo

SUMMARY:
This will be a multi-center, randomized, double-blind, placebo-controlled, crossover study to evaluate the effects of 2007/Fycompa (perampanel) on sleep, in subjects with well controlled partial onset seizures (on an antiepileptic drug [AED] monotherapy) who are experiencing sleep onset insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of epilepsy with partial onset seizures with or without secondary generalization, according to the ILAE Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history, with chart confirmation of previous EEG that is consistent with localization-related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history).
2. Subjects will be well controlled (defined as less than 1 seizure every 28 days) for a period of at least 3 months on a current AED monotherapy (defined as a single AED taken for at least 28 days before Screening), and have no history of AED polytherapy.
3. Male or female subjects, at least 18 years and no more than 50 years of age at the time of informed consent
4. Body Mass Index of 18 to 30 kg/m2
5. Meets Diagnostic and Statistical Manual-5 criteria for Insomnia Disorder:

   1. Complains of dissatisfaction with nighttime sleep in the form of difficulty getting to sleep or difficulty staying asleep
   2. Frequency of complaint is at least 3 times per week
   3. Duration of complaint is at least 3 months
   4. Associated with complaint of daytime impairment
6. Confirmed problems with sleep onset insomnia as evidenced by response to "Time to Fall Asleep" question on the PSQI at Screening of at least 45 minutes
7. Confirmed problems with sleep onset insomnia as evidenced by habitual median sSOL of at least 45 minutes obtained from sleep diary responses for the last consecutive 7 days of the Screening/Baseline Period
8. Confirmed problems with sleep onset insomnia as evidenced by LPS of at least 20 minutes on the baseline PSG
9. Provide written informed consent, signed by the subject before entering the study or undergoing any study procedures
10. Willing and able to comply with all aspects of the protocol
11. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] or a human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
12. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
13. Females of childbearing potential must not participate in a conception process (ie, active attempt to become pregnant or to impregnate, in vitro fertilization) and must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia), for at least 4 weeks before dosing, throughout the entire study period and for 4 weeks after study drug discontinuation. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 4 weeks after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 4 weeks after study drug discontinuation.

Exclusion criteria

1. Hypersensitivity to any component of Fycompa
2. Subjects with other sleep problems (except for sleep onset or mixed sleep onset and sleep maintenance insomnia) based on history, standard sleep questionnaires, and PSG at Screening.
3. Subjects with a diagnosis of a sleep-related breathing disorder, apnea-hypopnea index of more than 15, periodic limb movement disorder of more than 15, restless legs syndrome, nightmare disorder, sleep terror disorder, sleepwalking disorder, REM behavior disorder, narcolepsy, or circadian rhythm sleep disorder.
4. Subjects with current evidence of unstable psychotic disorder, major depressive disorder, bipolar disorder, or generalized anxiety disorder based on a psychiatric interview at Screening, or subjects diagnosed with psychotic disorder or major depressive disorder within 2 years before Screening based on clinical history
5. Subjects on strong cytochrome P450 (CYP) 3A inducers other than AEDs (eg, rifampin, St. John's Wort)
6. Subjects on EIAEDs: carbamazepine, oxcarbazepine, and phenytoin or eslicarbazepine (presumed EIAED)
7. Using a prescription or over the counter medication for the purpose of treating sleep disturbance, including sedating antihistamines, within 14 days before dosing
8. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or planning to travel across more than 3 time zones during the study
9. Excessive caffeine use (defined as more than 4 cups of coffee a day, or its equivalent)
10. Shift workers, defined as subjects who typically start work hours after 16:00 (4 pm) or before 4:00 (4 am)
11. Any history of a medical condition or concomitant medical condition that in the opinion of the investigator(s) would compromise the subject's ability to safely complete the study, including significantly abnormal laboratory results or any physical or mental condition that prevents compliance with the protocol
12. Use of illegal recreational drugs or recent history (within 2 years before the Screening Visit) of alcohol or drug/solvent dependency or abuse or a positive screen for drugs of abuse using a standard Urine Drug Screen at Screening
13. A clinically significant electrocardiogram (ECG) abnormality, including a prolonged QT interval/corrected QT interval defined as more than 450 msec based on an ECG at Screening
14. Currently enrolled in another clinical study or participated in any clinical study with an investigational drug, biologic, or device within 1 month before Screening (Visit 1), or within approximately 5 half-lives of the previous investigational compound, whichever is longer
15. Previous use of perampanel or participated in previous perampanel studies
16. Any suicidal ideation with intent with or without a plan at Screening or Baseline or within 6 months before Screening (ie, answering 'Yes' to questions on the Suicidal Ideation section of the electronic version of the Columbia Suicide Severity Rating Scale [eC-SSRS])
17. Suicide attempt(s) within approximately the last 2 years or suicidal ideation within the last 6 months before the Screening visit (using the Suicidal Behavior Section of the eC-SSRS)
18. Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase and aspartate aminotransferase due to concomitant medication(s) will be allowed if they are less than 3 times the upper limit of normal
19. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the Investigator(s) could affect the subject's safety or interfere with the study assessments
20. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors
21. Presence of an implanted vagal nerve stimulator
22. Have had multiple drug allergies or a severe drug reaction to an AED, including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in latency to persistent sleep (LPS) using Polysomnography (PSG) | Baseline, week 5 and week 14

SECONDARY OUTCOMES:
Change from baseline in Sleep Efficiency (SE) using Polysomnography (PSG) | Baseline, week 5 and week 14
Change from baseline in Subjective Sleep onset Latency (SSOL) using Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 5 and week 14
Mean reciprocal reaction time on Psychomotor Vigilance Task (PVT) to assess sustained attention | Baseline, week 5 and week 14
Short delay and long delay verbal recall using Rey Auditory Verbal Learning Test (RAVLT) | Baseline, week 5 and week 14
Measure number of seizures using Seizure Diary | baseline up to 18 weeks
Measure severity of suicidal ideation and behavior by eC-SSRS Electronic version of the Columbia Suicide Severity Rating Scale | baseline up to 18 weeks
Safety and tolerability of Perampanel as a measure of Adverse Events/ Serious Adverse Events | baseline up to 18 weeks